CLINICAL TRIAL: NCT06137443
Title: Enhancing Balance and Mobility in Incomplete Spinal Cord Injury With an Overground Gait Trainer
Brief Title: Enhancing Balance and Mobility in Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-MSS-01
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injuries; Walking, Difficulty
MeSH Terms: conditions — Spinal Cord Injuries; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance Training (Experimental): The study included five participants who were over 18 years of age and had experienced a spinal injury within the past year. These participants were classified as AIS D (American Spinal Injury Association Impairment Scale). Patients underwent treatment for eight weeks, with walking and balance exercises on Andago performed three days a week. In addition, conventional in-bed exercises, including stretching, strengthening, and mobility exercises, were administered for 40 minutes, two days a week.
  Interventions: Device: Balance Training

INTERVENTIONS:
Device: Balance Training — Patients underwent treatment for eight weeks, with walking and balance exercises on Andago performed three days a week. In addition, conventional in-bed exercises, including stretching, strengthening, and mobility exercises, were administered for 40 minutes, two days a week.

SUMMARY:
The goal of this clinical trial is to compare the effects of balance therapy with an overground gait trainer in incomplete spinal cord injury (SCI). The main questions it aims to answer are:

* Is balance therapy with an overground gait trainer effective in improving functional ambulation in SCI?
* Is balance therapy with an overground gait trainer effective in enhancing Activities of Daily Living in SCI?

Participants treated with either:

• Overground gait trainer along with conventional exercise therapy

DETAILED DESCRIPTION:
Background: Spinal Cord Injury (SCI) and similar pathologies not only negatively affect a person's ability to walk but also have adverse effects on their participation in social, vocational, and recreational activities. The correction of walking impairments resulting from SCI is one of the most important goals of rehabilitation, as it is essential for a person's social and vocational integration. When considering balance function, the use of challenging balance and walking exercises at an adequate level is necessary to trigger motor learning. Ensuring the patient's safety is the primary priority when using advanced balance and walking exercises based on the patient's current condition. In this study, Andago V2.0 (Hocoma AG, Volketswil, Switzerland) has been preferred for ensuring safety by adapting to patient movements. The main objective of the study was to assess the impact of Andago on balance in patients with motor incomplete SCI. The secondary aim was to evaluate its influence on quality of life and independence. Methods: The study included five participants who were over 18 years of age and had experienced a spinal injury within the past year. These participants were classified as AIS D (American Spinal Injury Association Impairment Scale). Patients underwent eight-week treatment, with walking and balance exercises on Andago performed three days a week. In addition, conventional in-bed exercises, including stretching, strengthening, and mobility exercises, were administered for 40 minutes, two days a week. Modified Borg Scale (MBS), Ten-Meter Walking Test (10MWT), Timed Up and Go Test (TUG), Walking Index in Spinal Cord Injury II (WISCI II), Berg Balance Scale (BBS), Visual Analogue Scale (VAS) for fear of falling, Spinal Cord Independence Measure (SCIM III), World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) were used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injured below T4
* Time from injury < 1 year
* D level on AIS (American Spinal Injury Association Impairment Scale)
* Patients with spinal stabilization

Exclusion Criteria:

* Osteoporosis
* An implanted electronic device
* other neurological diseases
* Cardio-pulmonary diseases
* Orthopedic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 11 months
  Berg Balance Scale for balance assessment

SECONDARY OUTCOMES:
Ten-Meter Walking Test | 11 months
  Ten-Meter Walking Test for overground walking speed assessment
Timed Up and Go Test | 11 months
  Timed Up and Go Test overground walking assessment
Walking Index in Spinal Cord Injury II | 11 months
  Walking Index in Spinal Cord Injury II for walking independence level assessment
Modified Borg Scale | 11 months
  Modified Borg Scale for subjective fatigue assessment
Visual Analogue Scale | 11 months
  Visual Analogue Scale (VAS) for fear of falling assessment
Spinal Cord Independence Measure (SCIM III) | 11 months
  Spinal Cord Independence Measure (SCIM III) for activity of daily living assessment
World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) | 11 months
  World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) for quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu P, Zhang W, Liu Y, Sheng C, So KF, Zhou L, Zhu H. The effects and potential mechanisms of locomotor training on improvements of functional recovery after spinal cord injury. Int Rev Neurobiol. 2019;147:199-217. doi: 10.1016/bs.irn.2019.08.003. Epub 2019 Sep 16. PMID 31607355
- [Background] Hayta E, Elden H. Acute spinal cord injury: A review of pathophysiology and potential of non-steroidal anti-inflammatory drugs for pharmacological intervention. J Chem Neuroanat. 2018 Jan;87:25-31. doi: 10.1016/j.jchemneu.2017.08.001. Epub 2017 Aug 10. PMID 28803968
- [Background] Finlayson ML, Peterson EW. Falls, aging, and disability. Phys Med Rehabil Clin N Am. 2010 May;21(2):357-73. doi: 10.1016/j.pmr.2009.12.003. PMID 20494282
- [Background] Contreras-Vidal JL, A Bhagat N, Brantley J, Cruz-Garza JG, He Y, Manley Q, Nakagome S, Nathan K, Tan SH, Zhu F, Pons JL. Powered exoskeletons for bipedal locomotion after spinal cord injury. J Neural Eng. 2016 Jun;13(3):031001. doi: 10.1088/1741-2560/13/3/031001. Epub 2016 Apr 11. PMID 27064508
- [Background] Esquenazi A, Talaty M, Packel A, Saulino M. The ReWalk powered exoskeleton to restore ambulatory function to individuals with thoracic-level motor-complete spinal cord injury. Am J Phys Med Rehabil. 2012 Nov;91(11):911-21. doi: 10.1097/PHM.0b013e318269d9a3. PMID 23085703
- [Background] Fouad K, Tetzlaff W. Rehabilitative training and plasticity following spinal cord injury. Exp Neurol. 2012 May;235(1):91-9. doi: 10.1016/j.expneurol.2011.02.009. Epub 2011 Feb 17. PMID 21333646
- [Background] Leech KA, Kinnaird CR, Holleran CL, Kahn J, Hornby TG. Effects of Locomotor Exercise Intensity on Gait Performance in Individuals With Incomplete Spinal Cord Injury. Phys Ther. 2016 Dec;96(12):1919-1929. doi: 10.2522/ptj.20150646. Epub 2016 Jun 16. PMID 27313241